CLINICAL TRIAL: NCT00252226
Title: Quetiapine (Seroquel) Maintenance Treatment in Early Onset Bipolar Spectrum Disorders: An Open Prospective Longitudinal Study of the Effectiveness of Quetiapine Monotherapy in Preventing Relapse and Minimizing Neurocognitive Dysfunction Among Adolescents Manifesting Bipolar Spectrum Disorders
Brief Title: Quetiapine (Seroquel) Maintenance Treatment in Early Onset Bipolar Spectrum Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mood Disorders Center of Ottawa (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Paul Grof, MDCO
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: D1441L00024
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Bipolar Disorder
Keywords: Quetiapine; bipolar spectrum disorders
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
This is a single center, open prospective study to evaluate the effectiveness of quetiapine monotherapy in the maintenance treatment of adolescent patients with a bipolar spectrum disorder (bipolar I and bipolar II disorders, cyclothymia, and bipolar disorder not otherwise specified [bipolar NOS]) for a minimum of 48 weeks. Patients will be screened (enrolment phase) either when already stabilized or during an acute episode of mania/hypomania or depression.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent before initiation of any study-related procedures.
2. A lifetime diagnosis of bipolar spectrum disorder: bipolar I and bipolar II disorders, cyclothymia, bipolar NOS, as defined by the Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition (DSM-IV).
3. Male or female, between the ages of 12 and 20 years at enrolment.
4. No preventive treatment at least one month prior to enrolment.
5. Female patients of childbearing potential and who are sexually active must be using a reliable method of contraception. Reliable methods of contraception include hormonal contraceptives (e.g., oral contraceptive or long-term injectable or implantable hormonal contraceptive), double-barrier methods (e.g., condom and diaphragm, condom and foam, condom and sponge), intrauterine devices, and tubal ligation.
6. Able to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Known intolerance or lack of response to quetiapine fumarate as judged by the investigator.
2. Pregnancy or lactation. Female patients of childbearing potential must have a negative urine human chorionic gonadotropin (HCG) test at enrolment.
3. History of substance or alcohol dependence within three months of enrolment (except for caffeine or nicotine dependence), as defined by DSM-IV criteria.
4. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment.
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, and saquinavir. Should a new drug be started, investigators will consult the pharmacy as this list is not exhaustive.
6. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids.
7. Current use of fluvoxamine, nefazodone, or grapefruit juice.
8. Thyroid stimulating hormone (TSH) concentration outside of the normal range.
9. Unstable or inadequately treated medical illness (e.g., diabetes, angina pectoris, hypertension) as judged by the investigator.
10. History of hepatic disease, or elevated hepatic enzymes at entry testing.
11. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment.
12. Use of an experimental drug within 30 days of enrolment.
13. Previous trials of maintenance therapy.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Proportion of treated study patients maintained on monotherapy for the duration of the trial compared to the proportion requiring systematic adjunctive medication.

SECONDARY OUTCOMES:
Time to an episode recurrence (Montgomery-Asberg Depression Rating Scale
/Young Mania Rating Scale [MADRS/YMRS] > 15)
Time to hospitalization
Autobiographical Memory Interview (AMI) mean score over treatment
Clinical Global Impression-Bipolar Disorder (CGI-BP) score during treatment and at study completion
YMRS total score during treatment and at study completion
MADRS total score during treatment and at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Paul Grof, M.D., Principal Investigator — Mood Disorders Center of Ottawa; Anne Duffy, M.D., Principal Investigator — Mood Disorders Center of Ottawa
Locations (1):
- Mood Disorders Center of Ottawa, Ottawa, Ontario, Canada